CLINICAL TRIAL: NCT00897845
Title: Molecular Profiling of E2197 FFPE Samples Using a Custom 512 Breast Cancer Gene Set on the DASL Platform: Towards the Development of Predictive Gene Sets for Risk of Recurrence in Patients With Operable Breast Cancer Treated With Adjuvant Therapy
Brief Title: Studying Tumor Samples From Women Who Have Undergone Chemotherapy for Breast Cancer
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000598872; ECOG-E2197B-ICSC; E2197T2 (Other: ECOG-ACRIN Cancer Research Group)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Microarray Analysis; Immunohistochemistry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: RNA analysis
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tumor tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor samples from women who have undergone chemotherapy for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To identify gene sets for risk of recurrence using molecular profiling in samples from women with lymph node-positive or high-risk lymph node-negative breast cancer on clinical trial ECOG-E2197.

Secondary

* To define a set of significant genes as prognostic markers of recurrence.
* To compare the prognostic value of the Oncotype DX™ (ODX) 21 gene assay of clinical trial with gene sets determined in this study.
* To compare the DASL™ assay of the ODX 21 genes with ODX assay results of clinical trial.
* To compare the prognostic value of selected genes with gene sets determined in this study.

OUTLINE: This is a multicenter study.

Samples are used in molecular profiling by applying a custom panel of breast cancer-related genes to a cDNA-mediated Annealing, Selection, Extension, and Ligation (DASL™) assay, immunohistochemistry, and other studies.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer tumor samples collected on clinical trial ECOG-E2197
* Histologically lymph node-positive (N1-3) OR high-risk lymph node-negative disease
* Hormone receptor-positive or negative disease (status known)
* HER2 status known

PATIENT CHARACTERISTICS:

* Menopausal status not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples submitted for research from patients enrolled on E2197
Sampling Method: Non-Probability Sample
Enrollment: 2541 (Actual)
Dates: Start 2008-06-17 (Actual); Primary Completion 2013-12-02 (Actual); Study Completion 2013-12-02 (Actual)

PRIMARY OUTCOMES:
Correlation of results with Outcome | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Brian Leyland-Jones, MD, Study Chair — Emory University